CLINICAL TRIAL: NCT06840288
Title: Bronchoscopic Lung Ablation of Small Thoracic Tumors: the Blastt Registry
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1847; NCI-2025-01258 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Thoracic Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Small Thoracic Tumors

SUMMARY:
To aggregate, integrate, and analyze data facilitating the study of MD Anderson patients with a known diagnosis of lung cancer or metastases to the lungs who undergo robotic assisted bronchoscopic ablation of peripheral tumors.

DETAILED DESCRIPTION:
A. To aggregate, integrate, and analyze data facilitating the study of MD Anderson participants with a known diagnosis of lung cancer or metastases to the lungs who undergo robotic assisted bronchoscopic ablation of peripheral tumors.

B. To assess the intra-operative, peri-operative, and long-term safety outcomes of robotic assisted bronchoscopic ablation of peripheral lung tumors.

C. To evaluate different oncologic outcomes including local tumor progression (LTP) by RECIST criteria, local tumor progression free survival (LTPFS), progression free-survival (PFS), disease (cancer) specific survival (DSS), and overall survival (OS).

D. To provide a deeper understanding of the evolution of radiographic findings of bronchoscopically ablated lung tumors over time.

E. To evaluate tumor and participant-related risk factors that may be associated with safety (bleeding, pneumothorax, and local infection) and oncologic outcomes (LTPFS, PFS, DSS, and OS).

ELIGIBILITY:
Inclusion Criteria:

Patients with peripheral lung tumors (primary or metastatic) that have been or will be ablated via robotic bronchoscopy.

Exclusion Criteria:

Patients with planned bronchoscopic ablations of peripheral lung tumors that were aborted for technical reasons (ablation was not completed).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
To aggregate, integrate, and analyze data facilitating the study of MD Anderson patients with a known diagnosis of lung cancer or metastases to the lungs who undergo robotic assisted bronchoscopic ablation of peripheral tumors. | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F Casal, MD, Principal Investigator — Prinicipal Investigator
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT06840288/ICF_000.pdf